CLINICAL TRIAL: NCT06493526
Title: Safety of Calcineurin-Inhibitor Withdrawal in Zero-HLA DQ-Mismatched Kidney Transplant Recipients on a Concentration Controlled Mycophenolate Dose: A Prospective, Single Arm Pilot Study
Brief Title: Mycophenolate-Based Therapy for Kidney Transplant Recipients Without HLA-DQ Mismatch
Acronym: MyQURE
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Antwerp (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UZA-6402
Record Dates: First submitted 2024-06-18; First posted 2024-07-10 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-06

CONDITIONS: Kidney Transplantation
Keywords: mycophenolate mofetil; Calcineurin Inhibitor; calcineurin inhibitor withdrawal; HLA-DQ; rejection; area under the curve; withdrawal; pharmacokinetic; concentration-controlled; mismatches
MeSH Terms: conditions — Rejection, Psychology | interventions — Adrenal Cortex Hormones

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Withdrawal of calcineurin-inhibitors in zero-HLA DQ-mismatched kidney transplant recipients (Experimental): calcineurin-inhibitor withdrawal, continue on a concentration controlled mycophenolate dose (AUC12 target 60 h.mg/L)
  Interventions: Drug: Withdrawal of calcineurin-inhibitor, continue on concentration-controlled mycophenolate mofetil and corticosteroids.

INTERVENTIONS:
Drug: Withdrawal of calcineurin-inhibitor, continue on concentration-controlled mycophenolate mofetil and corticosteroids. — Mycophenolate mofetil dose will be optimized to an AUC12 of 60 h.mg/L, thereafter the calcineurin inhibitor will be withdrawn.

SUMMARY:
The goal of this clinical trial is to learn if calcineurin-inhibitor therapy (a drug commonly used to prevent rejection) can be safely stopped in kidney transplant recipients with a relatively low risk of rejection (being recipients of a first transplant, without any signs of pre-existing immunity against the graft, and having a good HLA match with the donor (no mismatch in HLA-DQ)). Before stopping the calcineurin-inhibitors, the remaining therapy with mycophenolate mofetil and corticosteroids will be optimized.The main questions it aims to answer are:

Is this approach safe, in terms of preventing rejection? Is this approach well tolerated? Will this approach lead to better kidney function and/or other beneficial effects?

DETAILED DESCRIPTION:
In summary, this pilot, prospective, single-arm open interventional study the investigators will include immune-quiescent zero-DQ mismatched kidney transplant recipients between 3-12 months post-transplant who are on a CNI-based regimen with corticosteroids and MMF. After optimization of MMF dose, targeted at an MPA AUC12 of 60 (±15) mg.h/L, CNIs will be tapered and stopped over a 4 week peri-od. Prednisolon dose will be temporarily increased to 10 mg/day at the day of CNI withdrawal for 14 days, and continued at 5 mg/d thereafter. The primary outcome is biopsy-proven rejection at 6 months after CNI withdrawal. Secondary outcomes will look at other markers of alloreactivity (dnD-SA without clinical or histological signs of rejection), tolerability of MMF in the defined range, infec-tious complications, and possible favorable effects of CNI withdrawal (on GFR, tubular function, blood pressure, lipid profile and diabetes).

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in this study, a subject must meet all of the following criteria:

* Adults ≥ 18 years old who received a first, zero-HLA-DQ mismatched kidney transplant between 3 and 12 months before screening. ((mis)matching based on the broad Eurotransplant Match determinant for DQA1 and on the split Eurotransplant Match determinant for DQB1
* Maintenance immunosuppressive therapy should consist of a calcineurin-inhibitor (tacrolimus or cyclosporine), MMF and corticosteroids
* subjects capable of giving informed consent
* eGFR ≥ 20 ml/min/1.73m² based on CKD-EPI Creatinine-Cystatin Equation at screening
* Recent HLA antibody testing (<6 weeks before screening)
* Absence of DSA (MFI > 500) at screening and in all historical samples
* Absence of subclinical rejection on a protocol kidney transplant biopsy according to latest Banff criteria (excl. borderline lesions)
* Recent assessment of CNI and MPA AUC (performed at least 8 weeks after transplantation, but <12 weeks before screening, )
* Recent OGTT in patients not on antidiabetic therapy (<3 months ago)

Exclusion Criteria:

* Receipt of a non-renal transplant
* HLA identical sibling donor transplant
* ABO incompatible kidney transplantation
* cdc-PRA at transplantation > 50%
* Ongoing treatment with immunosuppressive drugs other than CNI, MMF/MPA and cortico-steroids
* Prophylactic therapy with valganciclovir
* History of biopsy-proven acute rejection
* Unexplained rise in creatininemia >20% over the last 6 weeks
* Albuminuria > 1g/day ( based on latest 24h urine collection max 6 weeks ago)
* Chronic diarrhea or gastrointestinal disorders that interfere with the absorption or oral medi-cation
* Active peptic ulcer disease
* Active hepatitis B, hepatitis C or human immunodeficiency virus infection at the day of trans-plantation
* New diagnosis of malignancy since transplantation, except successfully treated nonmetastatic basal or squamous cell carcinoma of the skin
* Pregnancy or lactation
* Patients unwilling to use reliable anticonception during the study (Male patients or their untreated female partner must use reliable contraception during my-cophenolate treatment and for at least 90 days after stopping MMF treatment. Female patients who can get pregnant must use at least one reliable form of contraception before, during and for 6 weeks after stopping MMF treatment)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-08-20 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of biopsy proven rejection | at 26 weeks after CNI withdrawal
  Biopsy will be performed as clinically indicated, or in case DSA develop (directed against HLA -A, HLA-B, HLA-DR or HLA-DQ with a MFI > 500 and remaining present in a repeated test after 6 weeks (± 2 weeks)) to exclude subclinical rejection.

SECONDARY OUTCOMES:
Incidence of biopsy proven rejection | at 14 weeks and 1 year after CNI withdrawal
  Biopsy will be performed as clinically indicated, or in case DSA develop (directed against HLA -A, HLA-B, HLA-DR or HLA-DQ with a MFI > 500 and remaining present in a repeated test after 6 weeks (± 2 weeks)) to exclude subclinical rejection.
Incidence of de novo donor specific HLA antibodies (dnDSA) | at 14 weeks, 26 weeks and 1 year after CNI withdrawal
  • HLA antibody testing (Luminex SAB): at baseline (unless performed < 6 weeks ago), day 98, day 182, day 364 (and in case of suspected rejection)
Tolerability of MMF in the defined range | up to 1 year after CNI withdrawal
  Gastro-intestinal Symptom Rating Scale and Adverse events
Change in eGFR | Comparing day 0 (day of CNI withdrawal) to 14 weeks, 26 weeks and 1 year after CNI withdrawal
  eGFR (CKDepi-cystatine formula)
Change in creatinine clearance | Comparing day 0 (day of CNI withdrawal) to 14 weeks, 26 weeks and 1 year after CNI withdrawal
  24h creatinine clearance
Change in albuminuria | Comparing day 0 to 14 weeks, 26 weeks and 1 year after CNI withdrawal
  Albuminuria in mg/day
Change in albumin/creatinine ratio in urine | Comparing day 0 to 14 weeks, 26 weeks and 1 year after CNI withdrawal
  Albumine/creatinine ratio in urine
Change in beta-2 microglobulinuria | Comparing day 0 to 14 weeks, 26 weeks and 1 year after CNI withdrawal
  beta-2 microglobulinuria in mg/day
Change in beta-2 microglobulin/creatinine ratio in urine | Comparing day 0 to 14 weeks, 26 weeks and 1 year after CNI withdrawal
  beta-2 microglobuline/creatinine ratio in urine
Change in arterial hypertension | Comparing baseline to 1 year after CNI withdrawal
  Blood pressure in mmHg
Change in number of antihypertensive drugs | Comparing baseline to 1 year after CNI withdrawal
  number of antihypertensive drugs
Change in serum total cholesterol | Comparing baseline to 1 year after CNI withdrawal
  total cholesterol levels (mg/dl)
Change in serum LDL cholesterol | Comparing baseline to 1 year after CNI withdrawal
  LDL cholesterol levels (mg/dl)
Change in serum HDL cholesterol | Comparing baseline to 1 year after CNI withdrawal
  HDL cholesterol levels (mg/dl)
Change in serum fasting triglycerides | Comparing baseline to 1 year after CNI withdrawal
  fasting triglyceride levels (mg/dl)
Change in need for statin therapy | Comparing baseline to 1 year after CNI withdrawal
  type and dose of statin therapy
Change in HbA1C | Comparing baseline to 1 year after CNI withdrawal
  HbA1C (%)
Change in need for antidiabetic medication | Comparing baseline to 1 year after CNI withdrawal
  number and type of antidiabetic drugs
Change in fasting glucose levels | Comparing baseline to 1 year after CNI withdrawal
  fasting glucose level (mg/dL)
Change in body weight | Comparing baseline to 1 year after CNI withdrawal
  Body weight in kg

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Hellemans, MD PhD, Principal Investigator — Antwerp University Hospital, Department of Nephrology, Drie Eikenstraat 655, 2650 Edegem, BELGIUM; Hans de Fijter, MD PhD, Principal Investigator — Antwerp University Hospital, Department of Nephrology, Drie Eikenstraat 655, 2650 Edegem, BELGIUM
Locations (1):
- University Hospital Antwerp, Edegem, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: No